CLINICAL TRIAL: NCT05876585
Title: A Randomized, Double-Blinded, Placebo-Controlled, Phase III Clinical Trial to Investigate the Efficacy and Safety of Ondansetron (Danset - Adwia) Versus Placebo Plus the Standard of Care in the Treatment of Nausea and Vomiting in Adult Patients With Acute Gastroenteritis
Brief Title: Clinical Trial to Investigate the Efficacy and Safety of Ondansetron (Danset - Adwia) Versus Placebo Plus the Standard of Care in the Treatment of Nausea and Vomiting in Adult Patients With Acute Gastroenteritis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Genuine Research Center, Egypt (Industry)
Collaborators: Adwia Pharma, Egypt (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRC/ADGE/EG/38/III
Record Dates: First submitted 2023-03-22; First posted 2023-05-25 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Gastroenteritis
MeSH Terms: conditions — Gastroenteritis | interventions — Ondansetron; Metoclopramide

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized in a 1:1 allocation ratio to receive a single dose of ondansetron 8 mg injection (arm 1) or a single dose of metoclopramide 10 mg injection (arm 2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ondansetron 8 mg ampoule (Experimental): A clear, colorless, sterile solution for injection or infusion. Each 1 ml of the solution contains 2 mg of ondansetron as hydrochloride dihydrate.
  Interventions: Drug: Ondansetron 8 mg ampoule
- Metoclopramide 10 mg ampoule (Active Comparator): Metoclopramide 10 mg/ 2 ml solution for injection in ampoules. Each 2 ml of the solution contains 10 mg of metoclopramide hydrochloride equivalent to 10 mg of anhydrous metoclopramide
  Interventions: Drug: Metoclopramide 10 mg ampoule

INTERVENTIONS:
Drug: Ondansetron 8 mg ampoule — Study drug
  Other Names: Danset ampoule
  Arms: Ondansetron 8 mg ampoule
Drug: Metoclopramide 10 mg ampoule — Comparator drug
  Other Names: Primperan
  Arms: Metoclopramide 10 mg ampoule

SUMMARY:
A Randomized, Open-label, Active-Controlled Clinical Trial to Investigate the Efficacy and Safety of Ondansetron compared to Metoclopramide in the management of Nausea and Vomiting in Adult Patients with Acute Gastroenteritis.

DETAILED DESCRIPTION:
This is a phase III, randomized, open-label, active-controlled, two-arm, parallel-design, interventional clinical trial evaluating the efficacy and safety of ondansetron 8 mg IV/ IM injection compared to metoclopramide 10 mg in the management of nausea and vomiting in adult patients with acute gastroenteritis.

Study duration: 1 year for patients' enrollment and follow-up. Sample Size: 63 subjects per arm, 126 in total. Participants in the trial will be male and female patients aged between 18 and 65 years visiting the emergency room due to acute gastroenteritis.

Patients will be screened for eligibility and eligible patients will be randomized in a 1:1 allocation ratio to receive a single dose of ondansetron 8 mg injection (arm 1) or a single dose of metoclopramide 10 mg injection (arm 2). Randomization will be done using interactive web response technology.

After drug administration, the patients will be followed up for 24 hours, including at least 3 hours in the emergency room immediately after drug administration.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged between 18 and 65 years.
2. Patients diagnosed with acute gastroenteritis visiting the emergency room.
3. Patients considered by the attending physician to need an anti-emetic medication.
4. Patients able and willing to provide written informed consent.
5. Patients able and willing to complete the study procedures including compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Patients who received an anti-emetic medication during the past 24 hours.
3. History of hypersensitivity to any components of ondansetron or metoclopramide injection.
4. History of hypersensitivity to other selective 5HT3 receptor antagonists.
5. Patients with moderate or severe impairment of hepatic function.
6. Patients with moderate or severe renal impairment.
7. Patients with congenital long QT syndrome.
8. Patients who have or may develop prolongation of Qtc, including patients with electrolyte abnormalities, congestive heart failure, bradyarrhythmia, or patients taking other medicinal products that lead to QT prolongation or electrolyte imbalance.
9. Patients with hypokalemia or hypomagnesemia.
10. Patients with signs of subacute intestinal obstruction.
11. Patients currently using apomorphine hydrochloride.
12. Patients currently using levodopa or dopamine agonists.
13. Patients with gastrointestinal hemorrhage, mechanical obstruction, or gastrointestinal perforation.
14. Patients with a known history of neuroleptic- or metoclopramide-induced tardive dyskinesia.
15. Patients with epilepsy.
16. Patients with Parkinson's disease.
17. Patients with confirmed or suspected pheochromocytoma.
18. Patients with a known history of methemoglobinemia with metoclopramide or NADH-cytochrome b5 reductase deficiency.
19. Patients with a history of clinically-significant illness or any other major medical disorder that may interfere with subject treatment, assessment, or compliance with the protocol.
20. Patients with any chronic illness or prior treatment which in the opinion of the investigator should preclude participation in the trial.
21. Receipt of an investigational drug within 6 months prior to screening, or active enrolment in another investigational medication or device trial.
22. Inability to understand and cooperate with the investigators or to give valid consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients experiencing complete control of nausea and vomiting | 6 hours after receiving the study medication
  Measured by asking the patient hourly to assess their nausea and vomiting.
The proportion of patients experiencing complete control of nausea and vomiting | 24 hours after receiving the study medication
  Measured by asking the patient hourly to assess their nausea and vomiting.
The proportions of patients who experienced nausea, vomiting, or retching. | 6 hours hours after receiving the study medication
  Measured by asking the patient hourly to assess their nausea, vomiting, or retching.
The proportions of patients who experienced nausea, vomiting, or retching. | 24 hours after receiving the study medication
  Measured by asking the patient hourly to assess their nausea, vomiting, or retching.
The proportion of patients who needed intravenous rehydration | 24 hours after receiving the study medication
  Assessed as per physician's discretion
The proportion of patients who needed a rescue anti-emetic medication | 24 hours after receiving the study medication
  Assessed as per physician's discretion
The duration of stay at the emergency room before discharge | From date of admission until the date of discharge, up to 3 hours
  The duration from admission to discharge from the emergency room
Overall patient's and physician's satisfaction with the efficacy of the study medication | 24 hours after receiving the study medication
  Measured by asking the patient and the physician

SECONDARY OUTCOMES:
The number of adverse events and serious adverse events | 24 hours after receiving the study medication
  Comparison between the number of adverse events and serious adverse events reported in the ondansetron 8 mg group and the metoclopramide 10 mg group
Overall patient's satisfaction with the tolerability of the study medication | 24 hours after receiving the study medication
  Measured by asking the patient

CONTACTS AND LOCATIONS:
Overall Officials: Waleed El-Nabawy, MD, Ph.D, Principal Investigator — Department of Internal Medicine, Faculty of Medicine, Beni-Suef University, Beni-Suef, Egypt; Tarek Ibrahim, MD, Principal Investigator — Department of Internal Medicine, Faculty of Medicine, Fayoum University, Fayoum, Egypt; Ahmed Dabour, MD, Ph.D, Principal Investigator — Department of Internal Medicine, Faculty of Medicine, Benha University, Benha, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cardemil CV, Balachandran N, Kambhampati A, Grytdal S, Dahl RM, Rodriguez-Barradas MC, Vargas B, Beenhouwer DO, Evangelista KV, Marconi VC, Meagley KL, Brown ST, Perea A, Lucero-Obusan C, Holodniy M, Browne H, Gautam R, Bowen MD, Vinje J, Parashar UD, Hall AJ. Incidence, Etiology, and Severity of Acute Gastroenteritis Among Prospectively Enrolled Patients in 4 Veterans Affairs Hospitals and Outpatient Centers, 2016-2018. Clin Infect Dis. 2021 Nov 2;73(9):e2729-e2738. doi: 10.1093/cid/ciaa806. PMID 32584956
- [Background] Chow CM, Leung AK, Hon KL. Acute gastroenteritis: from guidelines to real life. Clin Exp Gastroenterol. 2010;3:97-112. doi: 10.2147/ceg.s6554. Epub 2010 Jul 15. PMID 21694853
- [Background] Diemunsch P, Conseiller C, Clyti N, Mamet JP. Ondansetron compared with metoclopramide in the treatment of established postoperative nausea and vomiting. The French Ondansetron Study Group. Br J Anaesth. 1997 Sep;79(3):322-6. doi: 10.1093/bja/79.3.322. PMID 9389849
- [Background] Domino KB, Anderson EA, Polissar NL, Posner KL. Comparative efficacy and safety of ondansetron, droperidol, and metoclopramide for preventing postoperative nausea and vomiting: a meta-analysis. Anesth Analg. 1999 Jun;88(6):1370-9. doi: 10.1097/00000539-199906000-00032. PMID 10357347
- See also: Stuempfig ND, Seroy J. Viral Gastroenteritis. [Updated 2022 Jun 21]. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2022 Jan — https://www.ncbi.nlm.nih.gov/books/NBK518995/